CLINICAL TRIAL: NCT04482192
Title: Continuous Paravertebral Block by Intraoperative Direct Access Versus Systemic Analgesia for Postthoracotomy Pain Relief
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Deebis, Professor cardiothoracic surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZU-IRB: 6289
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Post Thoracotomy Pain
Keywords: Paravertebral block; Postthoracotomy analgesia; Systemic analgesia; Lidocaine infusion
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic paravertebral block group (Active Comparator): Continuous thoracic paravertebral block with 1% lidocaine infusion for 3 postoperative days through a paravertebral catheter inserted intraoperatively by the surgeon.
  Interventions: Combination Product: Thoracic paravertebral block
- Systemic analgesia group (Active Comparator): patients in this group will receive paracetamol and ketorolac by intravenous infusion every 6 hours for 3 postoperative days
  Interventions: Drug: Systemic analgesia

INTERVENTIONS:
Combination Product: Thoracic paravertebral block — After ending pulmonary procedure, a pleural pouch created beside vertebral column, a catheter is inserted to the pouch for continuous infusion of 1% lidocaine for 3 postoperative days. Intravenous morphine sulfate (0.05mg/kg) was given as a rescue medication if the VAS ≥ 4.
  Other Names: Study group
  Arms: Thoracic paravertebral block group
Drug: Systemic analgesia — Systemic analgesia (SA) group receive 1gm paracetamol and 30 mg ketorolac by intravenous infusion every 6 hours for 3 days. Intravenous morphine sulfate (0.05mg/kg) was given as a rescue medication if the VAS ≥ 4.
  Other Names: Control group
  Arms: Systemic analgesia group

SUMMARY:
to evaluate the safety and efficacy of continuous paravertebral block by intraoperative direct access on postthoracotomy pain compared to systemic analgesia.

DETAILED DESCRIPTION:
Based on a pilot study of 20 participants, 10 in each group, the mean visual analogue score of pain at rest (VAS) ± Standard Deviation (SD) at 6 hours postoperatively for Thoracic paravertebral block group (TPVB) participants were 3.0 ± 1.4 and that for systemic analgesia (SA) participants were 4.2 ± 1.6. The calculated significant sample size with a power of 0.85 and alpha error of 0.05 was 60 participants, with 1:1 allocation in each group.

Eighty two participants were assessed for eligibility criteria to be included in the study, 18 participants were excluded pre-randomization, and one participant was excluded post-randomization due to re-exploration for bleeding. Sixty three participants were analyzed in the study. Thoracic paravertebral block group (TPVB group) included 32 participants and systemic analgesia group (SA group) included 31 participants.

Technique of intraoperative paravertebral catheter insertion:

The investigators used the technique that was described by Sabanathan et al in 1988[14] and modified by them in 1990 [15]. After completing the surgical pulmonary procedure and with the chest is still open, starting from the posterior end of the thoracotomy, parietal pleura is raised from the posterior chest wall to the vertebral body and for two spaces above and below the incision of thoracotomy creating a pouch. A 16-gauge disposable Tuohy needle is inserted percutaneously through a low posterior interspace. The needle is advanced until the tip appeared in the created pouch. The stylet is removed, and a 16-gauge side-holed epidural catheter is advanced into the created pouch and the needle is withdrawn. Using a curved forceps, a small defect is done in the extrapleural fascia to be directly in the paravertebral space. The cannula is passed to the paravertebral space through the defect and advanced cranially for 2 to 3 cm. The parietal pleura is reattached to the posterior edge of the wound and the catheter is secured. Then a bolus dose 15-20 ml of 1% lidocaine is injected through the catheter and the chest is closed as usual with one or two intercostal drainage tubes according to the surgical procedure.

Protocol of analgesia:

All participants, in both groups, received intravenous analgesia with 1gm paracetamol and 30 mg ketorolac half an hour before the end of surgery.

Systemic analgesia (SA) group continue to receive 1gm paracetamol and 30 mg ketorolac by intravenous infusion every 6 hours for 3 days. Thoracic paravertebral block (TPVB) group received continuous infusion of 0.1 ml/kg/h of 1.0% lidocaine (l mg/kg/h) using infusion pump through the inserted paravertebral catheter for 3 days. Intravenous morphine sulfate (0.05mg/kg) was given as a rescue medication if the VAS ≥ 4 for both groups. A senior nurse was responsible for handling the analgesia regimen and another nurse was responsible for recording pain score on visual analogue scale (VAS) and morphine consumption, as scheduled.

ELIGIBILITY:
Inclusion Criteria:

* • Elective posterolateral thoracotomy surgery

  * American Society of Anesthesiologists (ASA) physical status of II and III

Exclusion Criteria:

* • lack of patient consent.

  * patients younger than 18 years,
  * emergency surgery,
  * previous thoracotomy,
  * drug addiction,
  * allergy to paracetamol (acetaminophen) or ketorolac,
  * coagulopathy,
  * hepatic dysfunction,
  * chronic renal failure,
  * history of gastric ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Pain score on visual analogue scale (VAS) at rest | 24 hours after operation
  Paper-based visual analogue scale (VAS) is used for pain assessment. It provides a range of scores from 0-10. A higher score indicates greater pain intensity.
Pain score on visual analogue scale (VAS) on coughing | 24 hours after operation
  Paper-based visual analogue scale (VAS) is used for pain assessment. It provides a range of scores from 0-10. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Total morphine consumption | end of first postoperative day
  The summation of morphine consumption of the participant
Forced vital capacity (FVC) | 24 hours after operation
  measured by spirometer (Microspiro HI-298, Chest Corporation, Tokyo, Japan)
Forced expiratory volume in 1s (FEV1) | 24 hours after operation
  measured by spirometer (Microspiro HI-298, Chest Corporation, Tokyo, Japan)
Peak expiratory flow rate (PEFR) | 24 hours after operation
  measured by spirometer (Microspiro HI-298, Chest Corporation, Tokyo, Japan)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Deebis, MD, Principal Investigator — Zagazig University

IPD SHARING:
Plan to Share IPD: Yes
All authors of the study will share individual participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after ending total collection of data till ending of writing the manuscript
Access Criteria: personal communication

REFERENCES:
- [Result] Krakowski JC, Arora H. Con: Thoracic Epidural Block Is Not Superior to Paravertebral Blocks for Open Thoracic Surgery. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):1720-2. doi: 10.1053/j.jvca.2015.06.012. Epub 2015 Jun 10. No abstract available. PMID 26386503
- [Result] Fortier S, Hanna HA, Bernard A, Girard C. Comparison between systemic analgesia, continuous wound catheter analgesia and continuous thoracic paravertebral block: a randomised, controlled trial of postthoracotomy pain management. Eur J Anaesthesiol. 2012 Nov;29(11):524-30. doi: 10.1097/EJA.0b013e328357e5a1. PMID 22914044
- [Result] Sabanathan S, Smith PJ, Pradhan GN, Hashimi H, Eng JB, Mearns AJ. Continuous intercostal nerve block for pain relief after thoracotomy. Ann Thorac Surg. 1988 Oct;46(4):425-6. doi: 10.1016/s0003-4975(10)64657-7. PMID 3178353
- [Result] Berrisford RG, Sabanathan SS. Direct access to the paravertebral space at thoracotomy. Ann Thorac Surg. 1990 May;49(5):854. doi: 10.1016/0003-4975(90)90058-e. No abstract available. PMID 2339953
- [Result] Wojtys ME, Wasikowski J, Wojcik N, Wojcik J, Wasilewski P, Lisowski P, Grodzki T. Assessment of postoperative pain management and comparison of effectiveness of pain relief treatment involving paravertebral block and thoracic epidural analgesia in patients undergoing posterolateral thoracotomy. J Cardiothorac Surg. 2019 Apr 16;14(1):78. doi: 10.1186/s13019-019-0901-3. PMID 30992044
- [Result] Elia N, Lysakowski C, Tramer MR. Does multimodal analgesia with acetaminophen, nonsteroidal antiinflammatory drugs, or selective cyclooxygenase-2 inhibitors and patient-controlled analgesia morphine offer advantages over morphine alone? Meta-analyses of randomized trials. Anesthesiology. 2005 Dec;103(6):1296-304. doi: 10.1097/00000542-200512000-00025. PMID 16306743
- [Result] Batra RK, Krishnan K, Agarwal A. Paravertebral block. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):5-11. No abstract available. PMID 21804697
- [Result] Katayama T, Hirai S, Kobayashi R, Hamaishi M, Okada T, Mitsui N. Safety of the paravertebral block in patients ineligible for epidural block undergoing pulmonary resection. Gen Thorac Cardiovasc Surg. 2012 Dec;60(12):811-4. doi: 10.1007/s11748-012-0149-5. Epub 2012 Sep 16. PMID 22983833
- See also: Procedure specific postoperative pain management. (2015) Thoracotomy. — http://www.esraeurope.org/prospect